CLINICAL TRIAL: NCT02726542
Title: Augmenting Growth Hormone to Ameliorate Nonalcoholic Fatty Liver Disease in Adolescents
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Takara Stanley, Assistant Professor of Pediatrics, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2016p-000657
Record Dates: First submitted 2016-03-30; First posted 2016-04-01 (Estimated); Results first posted 2021-04-26 (Actual); Last update posted 2022-09-07 (Actual); Status verified 2022-08

CONDITIONS: NAFLD
Keywords: obesity; adolescence; fatty liver; growth hormone
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease; Obesity; Fatty Liver | interventions — Human Growth Hormone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Growth hormone (Experimental): Somatropin given by daily subcutaneous injection. Dose will begin at 1mg and be titrated based on insulin-like growth factor 1 (IGF-1) levels.
  Interventions: Drug: somatropin
- No treatment (No Intervention): (no study treatment - observation only)

INTERVENTIONS:
Drug: somatropin — Norditropin (growth hormone) given by injection using a pen-device
  Arms: Growth hormone

SUMMARY:
Fatty liver disease is an increasing problem in overweight and obese young adults. The purpose of this study is to test the effect of growth hormone on liver fat in obese young adults ages 18-29y with increased liver fat.

DETAILED DESCRIPTION:
Non-alcoholic fatty liver disease (NAFLD) is a significant health problem in obese adolescents. Obese children and adolescents have significant reductions in growth hormone secretion, and we hypothesize that augmenting growth hormone in this population will decrease liver fat. Growth hormone inhibits hepatic de novo lipogenesis, which is an important source of hepatic lipid. Patients with pituitary GH deficiency have a higher prevalence of NAFLD and non-alcoholic steatohepatitis (NASH) than the general population, and replacement of GH in these individuals reduces signs of liver damage. The purpose of this study is to test the hypothesis that growth hormone treatment will decrease liver fat quantity in young adults who begin the trial with more than 5% liver fat measured by magnetic resonance spectroscopy.

ELIGIBILITY:
Inclusion criteria:

1. Males and Females ages 18-29yo
2. BMI ≥95th percentile and/or ≥30kg/m^2
3. Hepatic fat ≥5% by hydrogen magnetic resonance spectroscopy (1H-MRS)
4. IGF-1 standard deviation score (SDS) < 0

Exclusion criteria:

1. Alcohol consumption of >14 drinks per week (Females) or >21 drinks per week (Males)
2. Use of insulin or oral anti-diabetic medications, or hemoglobin A1c (HbA1c) >7% or fasting glucose ≥126mg/dL
3. Use of corticosteroid, gonadal steroids, or methotrexate ≤ 3 months prior to baseline visit
4. Known diagnosis of alpha-1 antitrypsin deficiency, Wilson's disease, hemochromatosis, or autoimmune hepatitis
5. hemoglobin < 11.0 g/dL or weight < 50kg
6. aspartate aminotransferase (AST) or alanine aminotransferase (ALT) >2.5x upper limit of normal (ULN), total bilirubin > ULN, positive hepatitis B surface antigen (sAg), or positive hepatitis C antibody
7. Routine magnetic resonance imaging (MRI) exclusion criteria (including weight >450 pounds)
8. Use of weight-loss medications or previous weight loss surgery
9. Pregnant or breastfeeding, or, for sexually-active females, unwillingness to use an appropriate form of contraception during the study
10. Known cirrhosis or clinical evidence of cirrhosis or portal hypertension on imaging or exam
11. Use of growth hormone (GH) or growth hormone releasing hormone within the past 1 year
12. Change in lipid lowering or anti-hypertensive medications within 3 months of screening
13. Change in vitamin E or ursodiol <6 months before screen; subjects on stable doses of Vitamin E and/or Ursodiol for ≥6 months will be eligible.
14. History of malignancy or active malignancy
15. History of hypopituitarism, head irradiation or any other condition or chronic illness known to affect the GH axis

Ages: 18 Years to 29 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2017-05-03 (Actual); Primary Completion 2020-04-02 (Actual); Study Completion 2020-04-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Takara Stanley, MD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Growth Hormone | No Treatment
Started | 13 | 11
Completed | 10 | 10
Not Completed | 3 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Growth Hormone | No Treatment | Total
Number analyzed (Participants) | 13 | 11 | 24
Age, Continuous [Mean (Standard Deviation); unit: years] | 25 (3) | 23 (4) | 24 (4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 6 | 13
  Male | 6 | 5 | 11
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaskan Native | 1 | 0 | 1
  Asian | 1 | 1 | 2
  White | 9 | 6 | 15
  Other or more than 1 race | 2 | 4 | 6
  Hispanic (independent of race) | 4 | 4 | 8
Region of Enrollment [Number; unit: participants]
  United States | 13 | 11 | 24

OUTCOME MEASURES:

1. Primary Outcome: Change in Hepatic Fat Fraction
Description: change in hepatic fat fraction between baseline and 24 weeks as measured by hydrogen magnetic resonance spectroscopy
Time Frame: 24 weeks
Population: all available data used
Measure: Mean (Standard Deviation); unit: Percent (Hepatic fat fraction, percent)
Arm/Group | Growth Hormone | No Treatment
Number analyzed (Participants) | 9 | 9
Percent (Hepatic fat fraction, percent) | -3.0 (5.2) | 0.3 (3.5)

2. Secondary Outcome: Change in Aspartate Aminotransferase (AST)
Description: change in AST between baseline and 24 weeks
Time Frame: 24 weeks
Population: all available data used
Measure: Mean (Standard Deviation); unit: units per liter
Arm/Group | Growth Hormone | No Treatment
Number analyzed (Participants) | 10 | 10
units per liter | -3 (9) | -1 (4)

3. Secondary Outcome: Change in Alanine Aminotransferase (ALT)
Description: change in ALT between baseline and 24 weeks
Time Frame: 24 weeks
Population: all available data used
Measure: Mean (Standard Deviation); unit: units per liter
Arm/Group | Growth Hormone | No Treatment
Number analyzed (Participants) | 10 | 10
units per liter | -2 (9) | 1 (8)

4. Secondary Outcome: Change in Gamma Glutamyl Transferase (GGT)
Description: change in GGT between baseline and 24 weeks
Time Frame: 24 weeks
Population: all available data used
Measure: Mean (Standard Deviation); unit: units per liter
Arm/Group | Growth Hormone | No Treatment
Number analyzed (Participants) | 10 | 10
units per liter | -9 (30) | 5 (9)

5. Secondary Outcome: Change in Visceral Adipose Tissue
Description: Change in visceral adipose tissue cross-sectional area at the 4th lumbar vertebra as measured by magnetic resonance imaging between baseline and 24 weeks
Time Frame: 24 weeks
Population: all available data used
Measure: Mean (Standard Deviation); unit: square centimeters
Arm/Group | Growth Hormone | No Treatment
Number analyzed (Participants) | 9 | 9
square centimeters | -6 (50) | 6 (24)

ADVERSE EVENTS:
Time Frame: Adverse events were collected from participants while they were enrolled in the 6 month study period.
Description: Participants were asked about adverse events at every study visit. Of note, participants receiving GH were seen for 4 additional visits compared to those receiving no treatment in this open-label study, and thus had more visits at which adverse events were assessed.
Arm/Group | Growth Hormone | No Treatment
All-Cause Mortality (participants affected / at risk) | 0/13 | 0/11
Serious Adverse Events (participants affected / at risk) | 1/13 | 0/11
Other Adverse Events (participants affected / at risk) | 9/13 | 1/11
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Growth Hormone (N=13) | No Treatment (N=11)
Hospitalization (Surgical and medical procedures) | 1 (1) | 0 (0) — Hospitalization related to psychiatric issues (further description not available)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Growth Hormone (N=13) | No Treatment (N=11)
Headache transient (Nervous system disorders) | 4 (5) | 1 (1)
Injection Site Bruising (General disorders) | 4 (6) | 0 (0)
Upper Respiratory Tract Infection (Infections and infestations) | 2 (2) | 0 (0)
Acne (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Gingival hyperplasia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Acute allergic reaction (Immune system disorders) | 1 (1) | 0 (0) — Allergic reaction to intravenous arginine administration given as part of GH stimulation testing protocol
Tightness in Jaw (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Motor Vehicle Accident (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-07-31): https://cdn.clinicaltrials.gov/large-docs/42/NCT02726542/Prot_SAP_000.pdf